# Informed consent form and

# Authorization to use and disclose protected health information

Sponsor / Study Title: Division of Microbiology and Infectious Diseases (DMID) /

National Institute of Allergy and Infectious Diseases (NIAID), National Institute of Health(NIH) "A Phase 1, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics and Safety of Pretomanid in Participants with Renal Impairment Compared

to Participants with Normal Renal Function"

Protocol Number: 15-0037

**Principal Investigator:** 

(Study Doctor)

William Smith, M.D.

**Telephone:** 865-410-8300

865-305-9100 (24-Hour)

**Address:** Alliance for Multispecialty Research, LLC.

1928 Alcoa Highway, Suite 107

Knoxville, TN 37920

Alliance for Multispecialty Research, LLC. 1924 Alcoa Highway, 4 and 5 Northwest

Knoxville, TN 37920

Alliance for Multispecialty Research, LLC.

801 N. Weisgarber Road, Suite 100

Knoxville, TN 37909

## **Key information**

You are invited to take part in a research study. This research study is studying pretomanid as a possible treatment for highly drug-resistant tuberculosis in patients with varying degrees of kidney disease. NIH is paying for this research study.

This study is an open-label study. Open-label means that both you and your study doctor will know which study treatment you are receiving.

This study will have 2 parts: Part A and Part B. In Part A, we will enroll 6 healthy participants who will serve as controls in Group 1A and enroll 6 participants with severe kidney (renal) malfunction or impairment and End Stage Renal Disease (ESRD), but who are not on dialysis in Group 2. If the results from Part A show greater than or equal to 50% higher pretomanid in the

blood of participants in Group 2 relative to the controls in Group 1A and if there are no major safety concerns identified, then the study will continue with Part B.

In Part B, up to 24 more participants will be enrolled to investigate the
pharmacokinetics (PK) and safety in participants with mild or moderate renal
impairment. PK is the study of how your body absorbs, breaks down, and removes the
study drug from your body.

This study is planned to include a total of 36 male and female adult participants. The study will include 6 groups as follows:

#### Part A:

- Group 1A: 6 healthy participants (matched controls) with normal kidney function
- Group 2: 6 participants with severe renal impairment and end-stage renal disease who are not on dialysis

#### Part B:

- Group 1B: 6 healthy participants (matched controls) with normal kidney function
- Group 3: 6 participants with mild renal impairment
- Group 1C: 6 healthy participants (matched controls) with normal renal function
- Group 4: 6 participants with moderate renal impairment

Your study doctor will explain when and how to take the study drug. Each group will receive one single dose of study drug, in tablet form.

The group you are in will be selected based on your health status or renal impairment or disease.

Participants: Please read this form carefully. Take your time to ask the study doctor or study staff as many questions about the study as you would like. The study doctor or study staff can explain words or information that you do not understand. Reading this form and talking to the study doctor or study staff may help you decide whether to take part or not. If you decide to take part in this study, you must sign your name at the end of this form.

#### **Background and purpose**

You are being asked to participate in this research study because you have normal kidney (renal) function; mild, moderate, or severe impairment; or ESRD and are not on dialysis.

The purpose of this research study is to:

- Test the safety of the study drug, pretomanid.
- Measure the impact of mild, moderate, severe kidney (renal) impairment, or end-stage kidney disease in participants not requiring dialysis on the PK of pretomanid. PK is the study of how your body absorbs, breaks down, and removes the study drug from your body.

Pretomanid is a new drug developed to treat tuberculosis in adults who cannot be treated with other drugs. This form of the disease is called highly drug-resistant tuberculosis. Pretomanid is currently approved by the U.S. Food and Drug Agency (FDA) under a limited pathway to treat adults with highly resistant pulmonary tuberculosis.

The use of pretomanid in this study is investigational. Additional research on pretomanid, like this study, is intended to determine if the drug is safe and effective in people with kidney disease.

Because this is a study, pretomanid will only be given to you during this study and not after the study is over. Pretomanid may be called the "study drug" throughout this consent form.

About 36 participants will be in this study.

## What will happen during the study?

Your participation in this study will last approximately 92 days and will include approximately 6 study visits to the study center.

## Screening:

Before any study-related tests and procedures are performed, you will be asked to read and sign this consent document. The following screening tests and procedures will then be performed to determine if you qualify to take part in this study:

Visit 00A, First Screening Study Center (Day -28 to -7)

- Eligibility criteria will be reviewed and your demographic information (age, sex, race, ethnicity, birth date, etc.) will be recorded. All of the protocol inclusion criteria and none of the exclusion criteria should be met.
- Your medical and surgical history (including surgical sterilization) will be recorded, including history of alcohol and smoking status.
- Any prescription or nonprescription medications you have taken within the past 30 days will be documented.
- Your height and weight will be measured.
- Your vital signs will be measured, including oral temperature, sitting pulse rate and sitting blood pressure.
- A complete physical examination will be performed.
- An electrocardiogram (also known as ECG, it measures how your heart is beating) will be performed. Sticky patches will be applied to your chest and extremities. Male participants may need to shave some chest hair so that the patches will stick to their skin. Female participants may need to remove their bra.
- Biological samples will be collected. The following tests will be performed on your samples:
  - Routine clinical laboratory tests such as blood hematology and blood chemistry and liver function.
  - A blood test for estimated glomerular filtration rate (eGFR); this test measures your kidney function.

- O Blood tests for hepatitis B, hepatitis C, and HIV. If your test results show that you have hepatitis or HIV, the study doctor will notify the local state health agency to report your condition. The results of your test(s) will be disclosed (made known) to local health agencies as required by law. If needed, the study doctor will recommend treatment to you, or the study doctor or study staff member will refer you to your primary care provider. If you test positive for hepatitis or HIV infection, you will not be included in the study.
- You will be advised to not drink alcohol for at least 72 hours before admission.

## Visit 00B, Second Screen Study Center (Day -28 to -7)

- Your willingness to participate will be reconfirmed and documented prior to performing any further study procedures.
- A urine pregnancy test will be performed on participants of childbearing potential and must be negative to ensure eligibility.
- A urine drug and alcohol screen (by blood or breathalyzer) will be performed; the results
  will be kept with your study chart and will not be discarded. If you test positive and are
  not taking a valid prescription, you will not be included in the study. Opiates and
  benzodiazepines will not be allowed even if prescribed. Therefore, a blood sample will
  be collected for this purpose.

## Visit 00C, Study Center Admission, Day -1

- You will be admitted to the study center 12-24 hours before administration of the study drug.
- Participants will be reminded that they must fast overnight (i.e., at least 8 hours) prior to the administration of the study drug on Day 1
- Participant's willingness to participate will be reconfirmed and documented.
- Interim medical history will be reviewed and any changes since last visits will be noted.
- All concomitant medications will be reviewed with participants and any new concomitant medications taken since the screening visit will be reviewed with participants and assessed for continued eligibility.
- Eligibility criteria will be reviewed.
- Blood and urine samples will be collected. The following tests will be performed on your samples:
  - For participants of childbearing potential, a urine sample will be collected for a pregnancy test.
  - o A sample will be collected to screen for alcohol (by blood or breathalyzer).
  - A urine drug and alcohol screen will be performed; the results will be kept with your study chart and will not be discarded.
  - Alcohol and urine drug screen results will be checked when available.
     Participants with positive results who are not taking a valid prescription will be discharged. Opiates and benzodiazepines will not be allowed even if prescribed.
     Participants who are discharged because of a positive alcohol or urine drug screen will not be rescreened for enrollment.

- An intravenous (in the vein, IV) catheter may be placed during this visit or the next if needed for collection of blood samples.
- If you take medications at home, you will need to bring these with you to the study center (the study center will not provide your regular medications)

## **Study Treatment:**

Before, During and After administration of Study Drug, Day 1

- Eligibility criteria will be reviewed.
- Interim medical history, including an assessment for new medical conditions and stability of chronic diseases, will be obtained by interview of participants and any changes since the previous visit (Visit 00C) will be noted.
- Alcohol and urine drug screening results from Day -1 will be reviewed for participants
  whose alcohol and drug screening results were not previously available and who were
  not discharged on Day -1. Participants with positive results who not taking a valid
  prescription will be discharged. Opiates and benzodiazepines will not be allowed even if
  prescribed.
- Vital signs, including oral temperature, sitting pulse, and sitting blood pressure will be recorded.
- An intravenous (in the vein, IV) catheter may be placed during this visit if not placed during the previous visit.
- A targeted physical examination may be performed.
- Review of medications taken within the last 30 days
- Multiple blood and urine samples will be collected.
- A urine pregnancy test will be performed prior to administration of the study product on all women of childbearing potential. Results must be negative and known prior to receipt of the study product
- You will need to eat a high-fat, high-calorie breakfast (provided) 30 minutes
   ± 10 minutes before you take the study drug. You should eat this meal in about half an hour or less.
- You will take one dose of 200 mg pretomanid pill. A mouth check will be done.
- You cannot eat or drink for 2 hours after taking the pill.
- All adverse events (AEs)/ serious adverse events (SAEs) will be recorded.

## <u>After Study Treatment</u>:

Because this is a research study, the study drug will be given to you only during this study and not after the study is over.

Study Center Stay, Day 2 and Day 3.

- A targeted physical examination may be performed
- Your medical history and medications will be reviewed

- Vital signs, including oral temperature, sitting pulse, and sitting blood pressure will be recorded.
- Urine and blood samples will be collected
- If an intravenous catheter is placed, this will be removed (on Day 3)
- You will be given a urine collection container to take home with instructions (you must return the collected urine the next day (within 24 hours). You will be instructed to collect urine for 2 more days at home and keep urine container at room temperature with the cap on
- You will be allowed to go home after review by a study clinician after 48 hours. You may also remain at the study center through Visit 01N, if you and the study doctor prefer.
- All AEs/SAEs will be recorded.

## Visit 01M, Day 4, Study Center

You will return to the study center for a follow-up visit 3 days (72 Hours  $\pm$  4 Hours Post-dose) after the administration of the study drug. The following assessments will be performed at this follow-up visit or in the event you discontinue from the study early:

- Your medical history and medications will be reviewed
- A targeted physical examination may be performed.
- Vital signs.
- Your urine will be returned to clinic.
- A blood sample will be collected.
- Any side effects will be recorded.

**Important!** The urine that you collect at home must be returned to the clinic within 24 hours after the collection started.

## Visit 01N, Day 5, Study Center

You will return to the study center for a follow-up visit 4 days (96 Hours  $\pm$  4 Hours Post-dose) after the last dose of study drug. The following assessments will be performed at the follow-up visit or in the event you discontinue from the study early:

- Your medical history and medications will be reviewed
- A targeted physical examination may be performed
- Vital signs
- An ECG will be performed.
- Your urine PK sample will be collected at home in the provided urine containers and stored at room temperature for no more than 24 hours. This specimen will be returned to clinic at this visit and you will be provided with a new urine collection container. A blood sample for PK will be collected.
- A blood sample will be collected
- All AEs/SAEs will be recorded.

## Visit 02, Day 12±2 days, Study Center

You will return to the study center for a follow-up visit approximately 12 days after the administration of the study drug. The following assessments will be performed at the follow-up visit or in the event you discontinue from the study early:

- Your medical history and medications will be reviewed
- A targeted physical examination may be performed
- Vital signs
- For participants of childbearing potential, a urine sample will be collected for a pregnancy test.
- A blood sample will be collected
- All AEs/SAEs will be recorded.

#### Final Visit, Phone Call, Day 85 +7 days

- You will be asked if you or your partner became pregnant. If yes, we will ask for details
  about the pregnancy to report the pregnancy to the sponsor and to document the
  outcome of the pregnancy.
- All AEs/SAEs will be recorded.

## Early Termination Visit (If Needed)

The following activities will be performed at the early termination visit for participants who discontinue, are discontinued, or are terminated from the study early:

- Your medical history and medications will be reviewed
- A targeted physical examination may be performed. For participants with renal impairment, this targeted review of systems will also focus on renal disease and will include questions pertaining to changes in the frequency and volume of urine, requirement for dialysis, and mental status
- Vital signs, including oral temperature, sitting blood pressure, and sitting pulse will be obtained
- A blood sample may be collected
- All AEs/SAEs will be recorded
- Participants of childbearing potential will take a urine pregnancy test

#### **Expectations**

If you participate in this study, you will be expected to:

- Complete all required visits
- Tell the study doctor your full medical history.
- Tell the study doctor about any side effects, changes in health status, or new medical problems that arise during the study.
- Tell the study doctor if you (or your partner) become pregnant.

#### **Unscheduled Visit (if needed)**

Unscheduled visits will be allowed for the following reasons:

Management of AEs and SAEs.

- Performance of repeat or additional laboratory tests for clinically abnormal test values.
- For a repeat urine pregnancy test if the participant suspects pregnancy.
- Anytime the investigator believes that it is clinically appropriate for patient safety.

## Risks, side effects, and/or discomforts

We do not know all the possible side effects of the study drug. Like all medications, the study drug could cause side effects, although not everybody gets them. Most side effects are transient (temporary), mild to moderate. However, some people may experience serious side effects and may require treatment.

The following side effects have been experienced by people who took the study drug in single or multiple doses in Phase 1 studies of healthy participants:

## For pretomanid:

## Very common (greater than or equal to at least 1 in 10 people)

- Headache (approximately 3 in 10 or 31.5%)
- Nausea (approximately 1 in 10 or 11.8%)
- Anemia (approximately 1 in 10 or 10.7%)
- Rash (approximately 1 in 10 or 11.4%) (skin rash)

#### Other reported side effects for pretomanid include:

- Vomiting
- Transaminases increased (abnormal liver test which could indicate possible liver damage)

It is also possible that you could have side effects that we do not know about. You will be monitored for the duration of your time in the study. You should tell your study doctor about any changes in your health while taking part in the study.

#### **Allergic Reaction**

As with taking any drug, there is a risk of allergic reaction. If you have a very serious allergic reaction, you may be at risk of death. Some symptoms of allergic reactions are:

- Rash
- Wheezing and difficulty breathing
- Dizziness and fainting
- Swelling around the mouth, throat or eyes
- A fast pulse
- Sweating

Please seek treatment immediately and tell the study doctor and study staff if you have any of these symptoms.

## Risks of study procedures

- Blood samples: can cause faintness, inflammation of the vein, pain, bruising, or bleeding at the site of puncture. There is also a slight possibility of infection. A total of about 100 ml (less than ½ cup) of blood will be drawn during the study.
- Electrocardiogram (ECG): Skin irritation is rare but could happen during an ECG from the electrode adhesive
- Fasting: Fasting for up to 8 hours could cause dizziness, headache, stomach discomfort, or fainting

#### **Prohibited Medications**

Please review the medicines listed in the table below and tell the study staff if you are taking any of them.

| CYP3A (including 3A4) inhibitors and inducers | | | |
|---|---|---|---|
| Strong inhibitors | Moderate inhibitors | Strong inducers | Moderate inducers |
| <ul> <li>Posaconazole</li> </ul> | <ul> <li>Schisandra</li> </ul> | | |
| Ritonavir and | <ul> <li>Verapamil</li> </ul> | | |
| ritonavir- | | | |
| containing | | | |
| coformulations | | | |
| <ul> <li>Saquinavir</li> </ul> | | | |
| <ul> <li>Tucatinib</li> </ul> | | | |
| <ul> <li>Voriconazole</li> </ul> | | | |

CYP=cytochrome P450;

From https://www.uptodate.com/contents/image?imageKey=CARD%2F76992

#### **Unforeseen risks**

There may be unknown risks to a pregnancy, embryo, or fetus (unborn baby) if you or your female partner become pregnant.

If you experience any side effects or have any concerns, you should tell the study doctor or study staff immediately.

#### **Birth control restrictions**

Taking the study drug may involve risks to a pregnant participant, an embryo, fetus (unborn baby) or nursing infant. Therefore, if you are pregnant, planning to become pregnant, planning to father a child, or are breastfeeding a child, you cannot participate in this study.

Participants who are able to become pregnant (not sterilized via tubal ligation, bilateral oophorectomy, bilateral salpingectomy, hysterectomy, implanted contraceptive device placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year has passed since the last menses if menopausal):

To reduce the risk of pregnancy, you should use an effective method of birth control while you are participating in this study and for the duration of the study after the administration of the study drug. Acceptable methods of birth control for use in this study are the following:

- Not having sexual intercourse with men.
- Combined hormonal contraception this is a form of hormonal contraception that combines both an estrogen hormone and a progestogen hormone in varying forms: the pill, the patch, the vaginal ring, or an injection.
- Progestogen-only hormonal contraception this relies on progestogen hormones alone to prevent ovulation; there are several progestogen-only methods of contraception: pills, implants, injectables.
- Intrauterine devices a small often T-shaped birth control device that is inserted in the uterus.

- Intrauterine hormone-releasing system an intrauterine device that releases the hormone into the uterus.
- Bilateral tubal occlusion which means your fallopian tubes have been blocked.

The study doctor or study staff will discuss this with you.

If you become pregnant while you are participating in this study, tell your study doctor or study staff immediately. Your participation in this study will be ended. The study staff will follow your pregnancy to its outcome.

#### Men:

To reduce the risk of pregnancy, you should use an effective method of birth control while you are participating in this study and for the duration of the study. Acceptable methods of birth control for use in this study are the following:

- Not having sexual intercourse with women.
- Use of a barrier method (condom).
- Your female partner should use one of the following:
  - Combined hormonal contraception this is a form of hormonal contraception that combines both an estrogen hormone and a progestogen hormone in varying forms: the pill, the patch, the vaginal ring, or an injection.
  - Progestogen-only hormonal contraception this relies on progestogen hormones alone to prevent ovulation; there are several progestogen-only methods of contraception: pills, implants, and injectables.
  - o Intrauterine devices a small often T-shaped birth control device that is inserted in the uterus.
  - o Intrauterine hormone-releasing system an intrauterine device that releases the hormone into the uterus.
  - Bilateral tubal occlusion which means your fallopian tubes have been blocked.
- Vasectomy (male sterilization).

Semen donation is not allowed for the duration of the study.

The study doctor or study staff will discuss this with you.

If your female partner becomes pregnant while you are participating in this study, tell your study doctor or study staff immediately. She may be asked to provide consent to follow the pregnancy.

# Alternatives to participation

This research study is for research purposes only. The only alternative is to not participate in this study.

#### **New findings**

Any new important information that is discovered during the study and which may influence your willingness to continue participation in the study will be provided to you.

#### Benefits

This study is for research purposes only. There is no direct benefit to you from your participation in the study. Information learned from the study may help other people in the future.

## **Compensation for participation**

You will be paid if you complete this study. You will be paid for the visits you complete according to the following schedule:

- \$150.00 for the completed screening visit.
- \$425.00 for the completion of study Days -1, 1, 2, 3, 4 and 5.
- \$50.00 for the completion of study Day 12.
- \$200.00 for the completion of study Day 85.

You will be paid following each completed study visit. If you do not complete the study, for any reason, you will be paid for each study visit you do complete.

If you decide to leave the study early, you will be paid \$150.00 for the completion of the early termination visit.

• \$150.00 for the completion of unscheduled visits.

If you have any questions regarding your compensation for participation, please contact the study staff.

## Confidentiality

Records of your participation in this study will be held confidential except when sharing the information is required by law or as described in this informed consent. The study doctor, the sponsor or persons working on behalf of the sponsor, and under certain circumstances, the U.S. FDA and the Institutional Review Board (IRB) will be able to inspect and copy confidential study-related records which identify you by name. This means that absolute confidentiality cannot be guaranteed. If the results of this study are published or presented at meetings, you will not be identified.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

To make sure that the health information collected in this study is accurate, it will need to be checked from time to time against your medical records. Some persons may need to see these records in order to monitor the research and verify the accuracy of the study data, including:

- A limited number of representatives from the study sponsoring drug company (namely its monitors and auditors),
- The research ethics review board Advarra IRB (an independent ethics committee that reviewed the ethical aspects of this study to help protect the rights and welfare of study participants),
- Government regulatory authorities including Health Canada, the U.S. FDA and other foreign regulatory agencies.

Your study records including confidential information about you collected during the study will be kept at a secure location.

While every effort will be made to protect the privacy of your information, absolute confidentiality cannot be guaranteed. This does not limit the duty of the researchers and others to protect your privacy.

By signing this information and consent form, you consent to the collection, access, use and disclosure of your information as described above.

# **Certificate of confidentiality**

To help us protect your privacy, we have a Certificate of Confidentiality from the NIH. Study staff cannot provide to any person not connected with the research your name, or any materials that contain identifiable, sensitive information about you, unless permitted by a legal exception, such as state laws that require reporting of some contagious diseases. The most important protection provided by the Certificate is that the study staff cannot be forced to provide any of your identifiable, sensitive information, in any Federal, State, or local civil, criminal, administrative, legislative, or other proceeding, such as if there is a court subpoena, without your permission.

The study team will use the Certificate to resist any demands for information that would identify you.

Your information protected by the Certificate may still be disclosed or used when the information:

- 1. Is disclosed to people connected with the research; for example, information may be used for auditing or program evaluation internally by the NIH; or
- 2. Is required to be disclosed by Federal, State, or local laws, for example, when information must be disclosed to meet the legal requirements of the U.S. FDA. This does not include disclosure for use during legal proceedings as noted above;
- 3. Is necessary for your medical treatment and you have consented to this disclosure;
- 4. Is for other scientific research as allowed by applicable federal regulations;
- 5. Is disclosed with your consent.

The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing and dating below you consent to those disclosures.

## **Compensation for injury**

If you become ill or are injured while you are in the study, get the medical care that you need right away. You should inform the healthcare professional treating you that you are participating in this study. If you tell the study staff that you think you have been injured, then they will help you get the care you need.

If you are injured because of taking the study drug(s) or from procedures done for the purpose of this study, the insurance procured by ICON will cover those medical expenses necessary to treat your injury that are not paid by your medical insurance or any other third-party coverage. No long-term medical care or financial compensation for research related injuries will be provided by the NIH or the Federal government. By signing this document, you will not lose any of your legal rights or release anyone involved in the research from responsibility for mistakes.

To pay medical expenses, ICON will request to know some information about you like your name, date of birth, and Medicare Beneficiary Identifier (MBI). This is because ICON must check to see if you receive Medicare and if you do, report the payment it makes to Medicare.

#### Costs

There will be no charge to you for your participation in this study. The study drug, study-related procedures, and study visits will be provided at no charge to you or your insurance company.

#### **Future research studies**

Your private information or biospecimens collected during this study **will not be used or distributed for future research studies,** even if identifiers are removed.

#### **Commercial profit**

Your biospecimens collected during this study may be used for commercial profit (even if identifiers are removed) and **you will not share in this profit**.

#### **Genome sequencing**

There will be no genetic testing done with your samples in this study.

## Whom to contact about this study

During the study, if you experience any medical problems, suffer a research-related injury, or have questions, concerns, or complaints about the study such as:

- Whom to contact in the case of a research-related injury or illness;
- Payment or compensation for being in the study, if any;
- Your responsibilities as a research participant;

- Eligibility to participate in the study;
- The study doctor's or study site's decision to withdraw you from participation;
- Results of tests and/or procedures;

# <u>Please contact the study doctor at the telephone number listed on the first page of this consent document.</u>

If you seek emergency care, or hospitalization is required, alert the treating physician that you are participating in this research study.

An IRB is an independent committee established to help protect the rights of research participants. If you have any questions about your rights as a research participant, contact:

#### By <u>mail</u>:

Study Subject Adviser Advarra IRB 6100 Merriweather Dr., Suite 600 Columbia, MD 21044

or call **toll free**: 877-992-4724

or by **email**: <u>adviser@advarra.com</u>

Please reference the following number when contacting the Study Subject Adviser: <u>Pro00074582</u>.

## Voluntary participation / withdrawal

Your decision to participate in this study is voluntary. You may choose to not participate, or you may withdraw from the study for any reason without penalty or loss of benefits to which you are otherwise entitled and without any effect on your future medical care. However, please note that the U.S. FDA requires that any information collected up to the point of your withdrawal cannot be removed from the study.

The study doctor or the sponsor can stop your participation at any time without your consent for the following reasons:

- If it appears to be medically harmful to you;
- If you fail to follow directions for participating in the study;
- If it is discovered that you do not meet the study requirements;
- If the study is canceled; or
- For administrative reasons.

If you leave the study for any reason, the study doctor may ask you to have some end-of-study tests for your safety.

| l<br>o | | or or primary h | <b>n</b> health care provider notified by the study sit ificant findings related to my health (please | :e |
|---|---|---|---|---|
| | □ <b>Yes</b> (If yes, please complete the □ <b>No</b> | information be | pelow) | |
| N | Name and address of family doctor or primary health care | Name: | | |
| | | Address: | | |
| | provider: | | | |
| | Telephone and Fax Number: | Tel: | | |
| | · | Fax: | | |
| v<br>le | oluntarily agree to participate in t | this study until | ns have been answered to my satisfaction. I<br>il I decide otherwise. I do not give up any of r<br>will receive a copy of this signed consent | ny |
| P | articipant's Printed Name | | _ | |
| Participant's Signature | | | <br>Date | |
| | rinted Name of the Person Condu<br>Consent Discussion | icting the | _ | |

**Consent Discussion** 

Signature of the Person Conducting the

Date

# Witness signature for participants who cannot read

The study participant has indicated that he/she is unable to read. The consent document has been read to the participant by a member of the study staff, discussed with the participant by a member of the study staff, and the participant has been given an opportunity to ask questions of the study staff.

| Printed Name of Impartial Witness | |
|-----------------------------------|----------|
| Signature of Impartial Witness | <br>Date |

# Authorization to use and disclose protected health information

Health data may come from your study records or from existing records kept by your doctor or other health care workers.

For this study, the study staff may share health data about you with authorized users. Authorized users may include:

- Representatives of DMID.
- Representatives of ICON.
- Representatives of Advarra IRB (an Institutional Review Board that reviews this study).
- The U.S. Food and Drug Administration (FDA) and other US federal and state agencies.
- Government agencies to whom certain diseases (like HIV, hepatitis, and sexually transmitted diseases [STDs]) must be reported.
- Governmental agencies of other countries.
- Outside individuals and companies, such as laboratories and data storage companies, that work with the researchers and sponsor and need to access your information to conduct this study.
- Other research doctors and medical centers participating in this study, if applicable.
- Safety monitoring committee which oversees this study.

Your health data will be used to conduct and oversee the research, including for instance:

- To see if pretomanid works and is safe.
- For other research activities related to pretomanid

Once your health data has been shared with authorized users, it may no longer be protected by federal privacy law and could possibly be used or disclosed in ways other than those listed here.

Your permission to use and share health data about you will end in 50 years unless you revoke it (take it back) sooner.

You may revoke (take back) your permission to use and share health data about you at any time by writing to the study doctor at the address listed on the first page of this form. If you do this, you will not be able to stay in this study. No new health data that identifies you will be gathered after your written request is received. However, health data about you that has already been gathered may still be used and given to others as described in this form.

Your right to access your health data in the study records will be suspended during the study to keep from changing the study results. When the study is over, you can access your study health data.

If you decide not to sign this form, you will not be able to take part in the study.

#### Statement of authorization

I have read this form and its contents were explained. My questions have been answered. I voluntarily agree to allow study staff to collect, use and share my health data as specified in this form. I will receive a signed and dated copy of this form for my records. I am not giving up any of my legal rights by signing this form.

| Printed Name of Participant | |
|---|---|
| Signature of Participant | <br>Date |
| has been read to the participant by a memb | nnot read<br>/she is unable to read. This Authorization documen<br>per of the study staff, discussed with the participan<br>rticipant has been given an opportunity to ask |
| Printed Name of Impartial Witness | <u>-</u> |
| Signature of Impartial Witness | <br>Date |